CLINICAL TRIAL: NCT05502302
Title: App-Assisted Day Reconstruction to Reduce Treatment Burden and Logistic Toxicity in Cancer Patients
Brief Title: App-Assisted Day Reconstruction to Reduce Logistic Toxicity in Cancer
Status: Completed | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2022LS036; R41CA271962 (NIH)
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The number of new cases of cancer diagnosed in the U.S. was 1.7 million in 2017 and is expected to increase by 35% to 2.3 million in 2030[1]. Cancer treatments often create numerous logistic challenges in prioritizing and managing treatment and everyday life priorities and how these challenges affect their everyday lives and well-being (hence "logistic toxicity"). However, there are no established reliable tools to monitor patients' logistic challenges and the associated impacts; and logistic toxicity has been largely unaddressed in cancer care delivery. The objective is to develop the first digital health app for cancer patients to continuously monitor logistic toxicity in their daily lives. The app will combine objective data from mobile sensing with subjective self-reported data to form an app-assisted day reconstruction system that captures activity engagement and well-being information associated with cancer treatment-related activities and trips throughout the day.

DETAILED DESCRIPTION:
The proposed patient monitoring app that captures logistic toxicity information on an ongoing basis will empower patients to advocate for care that better fits their life, give providers new insights into potential reasons for treatment non-adherence and nonresponse, and allow health systems to design more patient-centered care regimens.

A participatory design approach will be used to inform the design of our system, performing in-depth interviews and follow-up surveys with 20 diverse patients undergoing treatment for cancer. Patients will supply examples of logistic toxicity and how they would like to measure and communicate logistic toxicity across scenarios. Follow-up surveys will ask participants to provide satisfaction ratings towards user interface sketches and app function narratives.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, currently receiving treatment for cancer, able to read/write/speak in English, and able to provide voluntary informed consent.

Exclusion Criteria:

* Those who are currently incarcerated or have opted out of research contact within M Health Fairview system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MHealth Fairview Cancer Clinics
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel I Vogel, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Masonic Cancer Center - University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cancer Patients: Patients will supply examples of logistic toxicity and how they would like to measure and communicate logistic toxicity across scenarios.
Period: Overall Study
Arm/Group | Cancer Patients
Started | 23
Completed | 15
Not Completed | 8
Not completed — Lost to Follow-up | 6
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cancer Patients
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Interviews
Description: Number of Interviews completed to help identify themes to develop a cancer-specific, multi-tiered activity/trip classification system to organize cancer treatment-related activities and trips in the app; and user stories to describe what the users want to do with the proposed app. 45-minute interviews.
Time Frame: 7 months
Measure: Number; unit: Interviews
Arm/Group | Cancer Patients
Number analyzed (Participants) | 23
Interviews | 20

2. Primary Outcome: Satisfaction Score Follow-Up Survey
Description: Participants with overall satisfaction with proposed system design will be measured using a 5-point Likert scale from not at all satisfied to very satisfied. The primary endpoint will be the proportion of participants who report an overall satisfaction score of 4.0 or above. 10-Minutes.
Time Frame: 7 months
Measure: Number; unit: Percentage of participants
Arm/Group | Cancer Patients
Number analyzed (Participants) | 15
Percentage of participants | 80

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Cancer Patients
All-Cause Mortality (participants affected / at risk) | 2/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT05502302/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT05502302/ICF_001.pdf